CLINICAL TRIAL: NCT07071493
Title: An Exploratory Preliminary Study on the Effect of Combined Transcranial Photobiomodulation(tPBM)-Transauricular Vagus Nerve Stimulation(taVNS) on Alcohol Craving and Neurophysiological Marker in Drinkers (in South Korea)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A-STEAM-2024-01; RS-2024-00420674 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2025-06-25; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Normal Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three Group Intervention Studies (Experimental): * Stimulation Program (5 Weeks) Each participant will follow one of the following programs, assigned randomly, five days a week for a total duration of five weeks.
  1. tPBM Group: Participants will receive transcranial photobiomodulation (tPBM) for 15 minutes per day.
  2. taVNS Group: Participants will receive transcutaneous auricular vagus nerve stimulation (taVNS) for 15 minutes per day.
  3. Combined Treatment Group: Participants will simultaneously receive both tPBM and taVNS for 15 minutes per day.
  Interventions: Device: tPBM Group, taVNS Group, Combined Treatment Group: Stimulation Program (5 Weeks)

INTERVENTIONS:
Device: tPBM Group, taVNS Group, Combined Treatment Group: Stimulation Program (5 Weeks) — Stimulation Program (5 Weeks) Each participant will follow one of the following programs, assigned randomly, five days a week for a total duration of five weeks.
  tPBM Group: Participants will receive transcranial photobiomodulation (tPBM) for 15 minutes per day.
  taVNS Group: Participants will receive transcutaneous auricular vagus nerve stimulation (taVNS) for 15 minutes per day.
  Combined Treatment Group: Participants will simultaneously receive both tPBM and taVNS for 15 minutes per day.

SUMMARY:
Study Summary This pilot study aims to explore the mechanisms and effects of non-invasive neurostimulation in individuals with alcohol use, in order to develop a more accessible and sustainable treatment approach for alcohol use disorder.

Objectives

To evaluate the impact of:

Transcranial photobiomodulation (tPBM) Transcutaneous auricular vagus nerve stimulation (taVNS) Combined tPBM + taVNS on alcohol craving and neurophysiological indicators.

Method Participants: 60 adults (30 at Severance Hospital, 30 at Samsung Medical Center) Design: Randomized into 3 groups (tPBM, taVNS, combined) Intervention: 15 minutes/day, 5 days/week for 5 weeks (home-based) Assessments: Questionnaires, neurocognitive tests, EEG, and heart rate variability (HRV) Safety: Weekly phone check-ins for monitoring adverse effects Follow-up: Post-intervention assessments after 5 weeks

ELIGIBILITY:
1) Inclusion Criteria

1. Adults aged between 19 and 40 years who are able to provide valid written informed consent.
2. Individuals who consume alcohol, have an AUDIT-K score of 4 or higher, and do not meet the DSM-5 criteria for alcohol use disorder.
3. Individuals who are capable of completing the 5-week stimulation program.
4. Individuals who voluntarily agree to participate and sign the informed consent form.

2) Exclusion Criteria

1. Individuals who cannot read or understand the informed consent (e.g., illiterate individuals, non-Korean speakers).
2. Individuals with impaired decision-making capacity.
3. Pregnant women.
4. Vulnerable populations, including individuals employed by or under the supervision of the research institution, investigators, or sponsors (e.g., employees, students, military personnel).
5. Individuals unable to comply with the 5-week stimulation protocol.
6. Individuals diagnosed with alcohol use disorder according to DSM-5 criteria.
7. Individuals diagnosed with a substance use disorder other than alcohol or nicotine.
8. Individuals with metal allergies that may interfere with EEG or stimulation devices.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Craving Measured by the Penn Alcohol Craving Scale (PACS) | Administered at baseline (V1), five weeks (V2)
  The Pennsylvania Alcohol Craving Scale (PACS) consists of 5 items, each rated on a scale from 0 to 6. The scale comprehensively assesses the frequency, intensity, and duration of alcohol craving, as well as the individual's ability to resist drinking. The total score ranges from 0 to 30, with a score of 20 or higher indicating a level consistent with a substance use disorder.
  To evaluate changes in alcohol craving before and after a 5-week brain stimulation intervention using the Penn Alcohol Craving Scale (PACS). The study will compare the change in craving scores across three groups: combined stimulation (tPBM+taVNS), tPBM-only, and taVNS-only.

SECONDARY OUTCOMES:
Change in EEG-Based Neurophysiological Markers | Administered at baseline (V1), five weeks (V2)
  To evaluate changes in EEG signals (e.g., power spectral density, event-related potentials) before and after 5 weeks of intervention.
Change in Heart Rate Variability (HRV) | Administered at baseline (V1), five weeks (V2)
  To assess autonomic nervous system changes through time-domain and frequency-domain HRV parameters.
Change in Alcohol Use Measured by Alcohol Use Disorders Identification Test (AUDIT) | Administered at baseline (V1), five weeks (V2)
  The AUDIT is a 10-item questionnaire designed to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Higher scores indicate more severe alcohol-related issues. A score of 8 or above suggests hazardous or harmful alcohol use. Score Range: 0-40
Change in Drinking Motives Measured by Drinking Motives Questionnaire-Revised (DMQ-R) | Administered at baseline (V1), five weeks (V2)
  The DMQ-R is a drinking motives scale developed to measure adult drinking motives. This tool consists of four subscales: enhancement motives, coping motives, conformity motives, and social motives, with a total of 20 items. Each drinking motive is assessed with 5 items, totaling 20 items overall, and each item is rated on a 5-point scale from 1 "Not at all" to 5 "Very much so." Higher scores in each drinking motive subscale indicate a stronger motivation for that particular type of drinking.
Change in Depressive Symptoms Measured by Beck Depression Inventory (BDI). | Administered at baseline (V1), five weeks (V2)
  The Beck Depression Inventory (BDI) is a self-report questionnaire developed based on clinical symptoms of depression to assess the severity of depressive symptoms across 21 areas, including emotional, cognitive, and motivational aspects. Each item is rated on a 4-point scale (0 to 3), with total scores ranging from 0 to 63. A total score of 0-9 indicates no depression, 10-23 indicates moderate depression, and a score of 24 or above indicates severe depression.
Change in Anxiety Symptoms Measured by Beck Anxiety Inventory (BAI). | Administered at baseline (V1), five weeks (V2)
  The Beck Anxiety Inventory (BAI) is a tool designed to measure the severity of anxiety, encompassing cognitive, emotional, and physical aspects of anxiety. It consists of 21 items. The BAI was primarily developed to distinguish anxiety from depression. Each item is rated on a 4-point scale (0 to 3), with total scores ranging from 0 to 63. A total score of 21 or below indicates minimal anxiety, 22-26 indicates moderate anxiety, 27-31 indicates severe anxiety, and a score of 32 or above indicates extreme anxiety.
Change in Sleep Quality Measured by Pittsburgh Sleep Quality Index (PSQI). | Administered at baseline (V1), five weeks (V2)
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses subjective sleep quality over the past month. It evaluates sleep quality across seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
Change in Impulsivity Measured by Barratt Impulsiveness Scale (BIS). | Administered at baseline (V1), five weeks (V2)
  The Korean version of the Barratt Impulsiveness Scale-11 (BIS-11) is one of the most widely used self-report questionnaires for measuring impulsivity. It consists of three subcomponents: cognitive impulsivity, motor impulsivity, and non-planning impulsivity. The scale includes 30 self-report items, including 11 reverse-scored items. Each item is rated on a 4-point Likert scale ranging from 1 ("Not at all true") to 4 ("Always true"). Scores are calculated by summing the items, taking into account the reverse-scored items. Higher total scores indicate greater impulsivity.
Change in readiness to change measured by the Korean version of the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES-K). | Administered at baseline (V1), five weeks (V2)
  The SOCRATES was originally designed to assess motivation for change in problem drinkers. The Korean version (SOCRATES-K) was adapted to better reflect the Korean context and is used to assess motivation for change in individuals with alcohol dependence or abuse. It consists of 19 items, each rated on a 5-point Likert scale ranging from 1 ("Not at all true") to 5 ("Always true").
Change in Interoceptive Awareness Measured by Multidimensional Assessment of Interoceptive Awareness (MAIA). | Administered at baseline (V1), five weeks (V2)
  The Korean version of the Multidimensional Assessment of Interoceptive Awareness (MAIA) is a self-report questionnaire that reflects recent approaches such as mindfulness and acceptance, focusing on how individuals relate to internal experiences, including bodily sensations. It consists of 32 items related to interoceptive awareness. Each item is rated on a 7-point Likert scale ranging from 0 ("Not at all true") to 6 ("Always true"). Higher total scores, calculated by summing item scores, indicate greater interoceptive awareness.
Change in Craving and Metacognitive Control Measured by Meta Cognitions Questionnaire (MCQ). | Administered at baseline (V1), five weeks (V2)
  The Korean version of the Metacognitions Questionnaire consists of 30 items and assesses metacognitive beliefs across five domains: positive beliefs about worry, negative beliefs about the uncontrollability and danger of worry, cognitive confidence, need to control thoughts, and cognitive self-consciousness. Each item is rated on a 4-point Likert scale ranging from 0 ("Do not agree") to 3 ("Strongly agree").
Change in Credit Assignment Task (CAT) | Administered at baseline (V1), five weeks (V2)
  Participants will choose between two options, with rewards delivered after variable and unpredictable temporal delays. This task assesses participants' learning strategy and ability to infer the causal relationship between actions and outcomes when feedback is delayed, probing their capacity for temporal credit assignment.
Change in Delay Discounting Task (DDT) | Administered at baseline (V1), five weeks (V2)
  Participants will complete a computer-based binary choice task in which they repeatedly choose between smaller immediate rewards and larger delayed rewards. The task is designed to assess delay discounting - the degree to which individuals devalue rewards as a function of delay.
Change in Loss Aversion Task (LAT) | Administered at baseline (V1), five weeks (V2)
  A binary choice procedure will be used to assess individual sensitivity to loss aversion, where participants choose between mixed gambles involving potential gains and losses versus a certain outcome. This task quantifies the relative weighting of losses compared to gains.
Change in Choice under Risk and Ambiguity Task (CRAT) | Administered at baseline (V1), five weeks (V2)
  A binary choice procedure will be conducted in which, on certain trials, the probability of winning will be hidden in order to assess decision making under ambiguity, as compared to decision making under risk.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Jung, Professor, MD, PhD, Principal Investigator — Department of Psychiatry, Yonsei University College of Medicine Severance Hospital, Yonsei University Health System
Locations (2):
- South Korea (2):
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No